CLINICAL TRIAL: NCT06762522
Title: Exploring Feasibility and Acceptability of Using Neurofeedback Interventions to Manage Cognitive, Affective and Behavioural Symptoms in Persons with Mild Cognitive Impairment
Brief Title: Exploring Feasibility, Acceptability and Impact of Using Neurofeedback with Persons with Mild Cognitive Impairment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Providence Health & Services (Other)
Responsible Party: Principal Investigator, Marian Luctkar-Flude, RN, PhD, Associate Professor, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 65459
Record Dates: First submitted 2024-06-11; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-10

CONDITIONS: Mild Cognitive Impairment
Keywords: Neurofeedback; Feasibility
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Cognitive Training; Control Groups

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Nonlinear dynamical neurofeedback (NLD) (Experimental): The NLD study intervention will consist of 10 sessions of NeurOptimal neurofeedback delivered twice a week over a 5-week period. The intervention will be delivered by a certified NeurOptimal trainer. The average session length is 45 minutes including setup. Additional time of 15-20 minutes will be required prior to sessions when the surveys are completed.
  Interventions: Other: Nonlinear dynamical neurofeedback (NLD)
- Low energy neurofeedback system (LENS) (Experimental): The LENS study intervention will consist of 5 sessions of LENS neurofeedback delivered by a certified LENS trainer once a week over a 5-week period. The average session length is 15 minutes including setup. Additional time of 15-20 minutes will be required prior to sessions when the surveys are completed.
  Interventions: Other: Low energy neurofeedback system (LENS)
- Brain Music (Experimental): The Brain Music study intervention will consist of a brain mapping data acquisition session to create the personalized music, followed by 5 weekly sessions to adjust the music that participants will listen to at home on a daily basis. Initial data acquisition and weekly sessions will take about 30 minutes. Additional time of 15-20 minutes will be required prior to sessions when the surveys are completed.
  Interventions: Other: Brain Music
- Usual Care (Other): The Usual Care control group will continue to be followed in the Memory clinic at intervals determined by their clinician. Participants will complete the pretest and post-test assessments and surveys at baseline and at the end of 5 weeks.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Nonlinear dynamical neurofeedback (NLD) — NeurOptimal nonlinear dynamical (NLD) neurofeedback brain training works as a detection and monitoring system of changes in cortical patterns within the brain, mirroring the brain activity that can be undermining optimal brain function, providing the brain with the information it needs to make its own adjustments which over time results in the brain functioning more efficiently and effectively. Two scalp sensors at C3 & C4 and two earclips at tops of ears (reference) and one on the earlobe (ground) are used to read EEG activity which is analyzed by the NeurOptimal software. As participants listen to music through earbuds, information is fed back to the individual by slight interruptions in the music. One session lasts 33.5 minutes.
  Other Names: NeurOptimal neurofeedback; Brain training
  Arms: Nonlinear dynamical neurofeedback (NLD)
Other: Low energy neurofeedback system (LENS) — Low energy neurofeedback system (LENS) therapy is an EEG-based direct neurofeedback system that stimulates the brain to reset itself and achieve optimal performance. Therapy consists of delivery of a tiny electromagnetic field carrying the feedback signal down the electrode wires for only one second at each of the chosen electrode sites during every session. Generally, between one and seven of the ordinary electrode sites are utilized during each session. Therapy is adapted to the participant's reactivity/sensitivity and the response of their nervous system.
  Other Names: Direct neurofeedback
  Arms: Low energy neurofeedback system (LENS)
Other: Brain Music — Chen Medimo Corp (CMC) Brain Music neurofeedback analyzes an individual's EEG brainwave patterns and translates them into orchestral music. Listening to this personalized brain music allows the individual to gain self-awareness and rewire and alter their own mental states. The Brain Music protocol requires regular in-person follow-ups for optimal results. Generally, the number of sessions varies based on individual needs and the progress made in response to the CMC Brain Music. A minimum of once a week in-person sessions is recommended for qEEG model updating to accurately track progress. Each session may last 30 minutes. Additionally, participants are advised to listen to their personalised music at least once a day, with a minimum of two listens per session. In general, participants may start to detect a change in their neurodevelopmental or cognitive function in 4-6 weeks.
  Other Names: Chen Medimo Corp. (CMC); CMC Brain Music
  Arms: Brain Music
Other: Usual Care — The Usual Care control group will be followed in the Memory clinic at intervals determined by their clinician. Usual Care for individuals with mild cognitive impairment (MCI) at the The Memory Clinic consists of inter-professional assessment, diagnosis and recommendations. There are currently no drugs approved to treat MCI. Therapy is aimed at managing treatable causes and contributors including medication side effects, thyroid problems, sleep apnea, vitabim B deficiency, depression, anxiety, and unrecognized or untreated difficulties with hearing or vision. Neurofeedback is not a component of the standard of care.
  Other Names: Control group
  Arms: Usual Care

SUMMARY:
The goal of this pilot study is to determine the feasibility, acceptability and potential impact of using neurofeedback interventions to manage cognitive, emotional, and behavioural symptoms in individuals with mild cognitive impairment (MCI). The main question[s] it aims to answer are: (1) What is the feasibility, acceptability, and appropriateness of using the Nonlinear Dynamical Neurofeedback intervention for persons living with MCI? (2) What is the feasibility, acceptability, and appropriateness of using the Low Energy Neurofeedback System (LENS) intervention for persons living with MCI? (3) What is the feasibility, acceptability, and appropriateness of using the Brain Music neurofeedback intervention for persons living with MCI? (4) What is the potential impact of five weeks of a neurofeedback intervention on cognitive, affective, and behavioural symptoms experienced by persons living with MCI? Participants will be randomly assigned to either the Nonlinear Dynamical (NLD), Low Energy Neurofeedback System (LENS), or Brain Music neurofeedback intervention groups or a control group receiving usual care.

DETAILED DESCRIPTION:
Mild cognitive impairment (MCI) involves more severe memory, language, thinking, or judgment problems than normal aging, often progressing to dementia. Current treatments, both pharmacological and non-pharmacological, show limited benefits, prompting the need for alternative approaches like neurofeedback. Neurofeedback is a non-invasive technique that enhances the central nervous system's flexibility and resilience, potentially boosting cognitive reserve and delaying cognitive decline. This study focuses on three advanced neurofeedback methods: Nonlinear Dynamical Neurofeedback (NLD), Low Energy Neurofeedback System (LENS), and Brain Music. Before conducting a full clinical trial, it's crucial to determine if these methods are feasible and acceptable for people with MCI. This pilot study aims to explore the feasibility, acceptability, and potential impact of using neurofeedback interventions to manage cognitive, emotional, and behavioural symptoms in individuals with mild cognitive impairment (MCI).

The study involves a quasi-experimental design with 20 participants recruited from the Providence Care Hospital Memory Clinic in Kingston, Ontario. Participants will be randomly assigned to either the NLD, LENS, or Brain Music intervention groups or a control group receiving usual care. Each intervention will last five weeks, with assessments conducted before and after the intervention period. Clinical outcomes measured include objective cognitive assessments using the Creyos Health Cognitive Assessment. Subjective self-reported measures will include the Short-Form Pittsburgh Sleep Quality Index (SF-PSQI) survey to measure sleep quality, the Beck Depression Inventory (BDI) to measure depressive symptoms, and the Beck Anxiety Inventory (BAI) to measure anxiety. Feasibility and acceptability will be evaluated based on participation rates, survey responses, and withdrawal rates, along with the resources needed for the study. Data analysis will involve repeated measures ANOVAs to identify trends and assess the reliability of the measures used, providing foundational data for future research on neurofeedback's efficacy in managing MCI symptoms This data will inform the design of a larger clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Adults with mild cognitive impairment (MCI) attending the Memory Clinic at Providence Care Hospital in Kingston, Ontario

Exclusion Criteria:

* Adults with cognitive issues related to a psychiatric diagnosis or acute brain injury

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-27 (Estimated); Primary Completion 2025-12-23 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility Measure 1: Study participation rates | Data will be collected throughout the study enrolment period of three months
  Feasibility of the neurofeedback interventions will be assessed by study participation rates.
Feasibility Measure 2: Survey response rates | Data will be collected throughout the study enrolment and delivery period of six months.
  Feasibility of the neurofeedback interventions will be assessed by survey response rates.
Feasibility Measure 3: Study withdrawal rates | Data will be collected throughout the study enrolment and delivery period of six months.
  Feasibility of the neurofeedback interventions will be assessed by study withdrawal rates.
Creyos Health Cognitive Assessment: Objective measure of cognition | Measurement will occur at three time points: (T0) at week 0, immediately before the first neurofeedback session, (T1) at week5, after the last neurofeedback session, and (T2) 5 weeks following the last neurofeedback session.
  The primary clinical outcome of cognition will be measured objectively using the Creyos Health Cognitive Assessment, an online platform of validated neurocognitive tasks and batteries that have been used in over 300 peer-reviewed studies to measure core elements of cognition. Individual raw scores on a task are compared with a population of individuals of the same gender and age group and presented as standard scores and percentiles and then adjusted to better reflect the individual's true cognitive ability. Scores are classified as average, below average or above average based on the standard score. We will use the 6-task version of the Creyos MCI battery as it appears to be adequate for monitoring and reduces testing time.
Feasibility Measure 4: Feasibility of Intervention Measure (FIM) | The FIM will be completed as part of the follow-up survey at T2, 5 weeks following the last neurofeedback session.
  Feasibility of the neurofeedback interventions will be assessed using the Feasibility of Intervention Measure (FIM) which is a subscale of The Triple P Tool. Scale items are scored on a Likert scale from 1 to 5 where higher scores indicate higher feasibility.
Feasibility Measure 5: Acceptability of Intervention Measure (AIM) | The AIM will be completed as part of the follow-up survey at T2, 5 weeks following the last neurofeedback session.
  Acceptability, of the neurofeedback interventions will be assessed using the Acceptability of Intervention Measure (AIM) which is a subscale of the Triple P Tool. Scale items are scored on a Likert scale from 1 to 5 where higher scores indicate higher acceptability of the intervention.
Feasibility Measure 6: Intervention Appropriateness Measure (IAM) | The IAM will be completed as part of the follow-up survey at T2, 5 weeks following the last neurofeedback session. Data will be collected throughout the study period of six months
  Appropriateness of the neurofeedback interventions will be assessed using the Intervention Appropriateness Measure (IAM) which is a subscale of the Triple P Tool. Scale items are scored on a Likert scale from 1 to 5 where higher scores indicate higher appropriateness of the intervention.

SECONDARY OUTCOMES:
Beck Anxiety Inventory: Anxiety | Measurement will occur at three time points: (T0) at week 0, immediately before the first neurofeedback session, (T1) at week 5, after the last neurofeedback session, and (T2) 5 weeks following the last neurofeedback session.
  The Beck Anxiety Inventory consists of 21 items to assess a broad range of emotional, physical, cognitive and behavioural symptoms that represent important dimensions of anxiety. The BAI shows high internal consistency (alpha=.92) and test-retest reliability over 1 week, r(81) = .75. Individual scale items are rated on a scale from 0 to 3. The total score is cauculted by finding the sum of the 21 items. Higher scores indicate higher levels of anxiety.
Beck Depression Inventory: Depression | Measurement will occur at three time points: (T0) at week 0, immediately before the first neurofeedback session, (T1) at week5, after the last neurofeedback session, and (T2) 5 weeks following the last neurofeedback session.
  The Beck Depression Inventory-II (BDI-II) consists of 21 items to assess the intensity of depression in clinical and normal patients over the preceding two weeks. Each item is a list of four statements arranged in increasing severity about a particular symptom of depression in alignment with the DSM-IV criteria. The BDI-II (Coefficient Alpha = .92) showed improved clinical sensitivity over the BDI (Coefficient Alpha = .86). ndividual scale items are rated on a scale from 0 to 3. The total score is cauculted by finding the sum of the 21 items. Higher scores indicate higher levels of depression.
Short-Form Pittsburgh Sleep Quality Index: Sleep quality | Measurement will occur at three time points: (T0) at week 0, immediately before the first neurofeedback session, (T1) at week5, after the last neurofeedback session, and (T2) 5 weeks following the last neurofeedback session.
  The Pittsburgh Sleep Quality Index (PSQI) assesses sleep quality over a 1-month time interval. Nineteen individual items generate 7 component scores and a global score. The PSQI demonstrates acceptable measures of internal homogeneity, consistency and validity, and distinguishes well between good and poor sleepers. We will use the short form SF-PSQI in this study, a 13-item scale that corresponds to 5 of the 7 components of the original tool. Total scores range from 0 to 21 with higher scores associated with poorer sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Marian Luctkar-Flude, PhD, Principal Investigator — Queen's University, School of Nursing
Locations (1):
- Providence Care Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
This is a small feasibility study, thus it will not be necessary to share any individual participant data with other researchers.

REFERENCES:
- [Background] Trambaiolli LR, Cassani R, Mehler DMA, Falk TH. Neurofeedback and the Aging Brain: A Systematic Review of Training Protocols for Dementia and Mild Cognitive Impairment. Front Aging Neurosci. 2021 Jun 9;13:682683. doi: 10.3389/fnagi.2021.682683. eCollection 2021. PMID 34177558
- [Background] Sitaram R, Ros T, Stoeckel L, Haller S, Scharnowski F, Lewis-Peacock J, Weiskopf N, Blefari ML, Rana M, Oblak E, Birbaumer N, Sulzer J. Author Correction: Closed-loop brain training: the science of neurofeedback. Nat Rev Neurosci. 2019 May;20(5):314. doi: 10.1038/s41583-019-0161-1. PMID 30911159
- [Background] Petersen RC, Lopez O, Armstrong MJ, Getchius TSD, Ganguli M, Gloss D, Gronseth GS, Marson D, Pringsheim T, Day GS, Sager M, Stevens J, Rae-Grant A. Practice guideline update summary: Mild cognitive impairment [RETIRED]: Report of the Guideline Development, Dissemination, and Implementation Subcommittee of the American Academy of Neurology. Neurology. 2018 Jan 16;90(3):126-135. doi: 10.1212/WNL.0000000000004826. Epub 2017 Dec 27. PMID 29282327
- [Background] McGirr A, Nathan S, Ghahremani M, Gill S, Smith EE, Ismail Z. Progression to Dementia or Reversion to Normal Cognition in Mild Cognitive Impairment as a Function of Late-Onset Neuropsychiatric Symptoms. Neurology. 2022 May 24;98(21):e2132-e2139. doi: 10.1212/WNL.0000000000200256. Epub 2022 Mar 29. PMID 35351783
- [Background] Gallagher D, Fischer CE, Iaboni A. Neuropsychiatric Symptoms in Mild Cognitive Impairment. Can J Psychiatry. 2017 Mar;62(3):161-169. doi: 10.1177/0706743716648296. PMID 28212495
- [Background] Alzheimer Society. (2024). Mild cognitive impairment. https://alzheimer.ca/en/about-dementia/other-types-dementia/conditions-related-dementia
- [Background] Beck AT, Epstein N, Brown G, Steer RA. An inventory for measuring clinical anxiety: psychometric properties. J Consult Clin Psychol. 1988 Dec;56(6):893-7. doi: 10.1037//0022-006x.56.6.893. No abstract available. PMID 3204199
- [Background] Beck, A.T., Steer, R.A., &amp; Brown, G.K. (1996). Beck Depression Inventory-II (BDI-II). https://www.pearsonassessments.com/store/usassessments/en/Store/Professional-Assessments/Personality-%26-Biopsychosocial/Beck-Depression-Inventory/p/100000159.html?tab=product-details
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Campos da Paz, V.K., &amp; Tomaz, C. (2020). Neurofeedback training on aging: Prospects on maintaining cognitive reserve. In K.F.Shad &amp; K.H. Dogan (Eds.) Neurological and mental disorders. http://dx.doi.org/10.5772/intechopen.90847
- [Background] Canadian Task Force on Preventive Health Care. (2023). Cognitive impairment: Clinician summary. https://canadiantaskforce.ca/cognitive-impairment-clinician-summary/
- [Background] Chen Medimo Corp. (2023). NeuroRecovery Training (NRT). https://chenmedimo.org/nrt
- [Background] Corbo I, Marselli G, Di Ciero V, Casagrande M. The Protective Role of Cognitive Reserve in Mild Cognitive Impairment: A Systematic Review. J Clin Med. 2023 Feb 22;12(5):1759. doi: 10.3390/jcm12051759. PMID 36902545
- [Background] Creyos, Canada. (2024). Creyos: Quickly gain validated and powerful brain health insights. https://creyos.com/
- [Background] Famodu OA, Barr ML, Holaskova I, Zhou W, Morrell JS, Colby SE, Olfert MD. Shortening of the Pittsburgh Sleep Quality Index Survey Using Factor Analysis. Sleep Disord. 2018 Apr 12;2018:9643937. doi: 10.1155/2018/9643937. eCollection 2018. PMID 29850262
- [Background] Fitzpatrick-Lewis D, Warren R, Ali MU, Sherifali D, Raina P. Treatment for mild cognitive impairment: a systematic review and meta-analysis. CMAJ Open. 2015 Dec 1;3(4):E419-27. doi: 10.9778/cmajo.20150057. eCollection 2015 Oct-Dec. PMID 26770964
- [Background] Fydrich, T., Dowdall, D., &amp; Chambless, D.L. (1992). Reliability and validity of the Beck Anxiety Inventory. Journal of Anxiety Disorders, 6(1), 55-61. https://doi.org/10.1016/0887-6185(92)90026-4
- [Background] Ochs, L. (2006). The low energy neurofeedback system (LENS): theory, background, and introduction. Journal of Neurotherapy, 10(2-3), 5-39. https://doi.org/10.1300/J184v10n02_02
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Zengar Institute Inc. (2024). NeurOptimal® Brain Training eBook. https://neuroptimal.com/discover-neuroptimal-ebook/